CLINICAL TRIAL: NCT05530330
Title: Markers of Platelet Activation foR Identification of Late Onset Sepsis in Preterm Infants
Acronym: PARENT
Status: Completed | Type: Observational
Sponsor: University College Dublin (Other)
Collaborators: The Rotunda Hospital (Other); National Maternity Hospital, Ireland (Other); Wellcome Trust (Other); Health Research Board, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: REC-2022-008
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-12

CONDITIONS: Late-Onset Neonatal Sepsis; Necrotising Enterocolitis; Culture Negative Neonatal Sepsis
Keywords: Sepsis; Neonatal; Preterm
MeSH Terms: conditions — Neonatal Sepsis; Enterocolitis, Necrotizing; Sepsis; Premature Birth | interventions — Platelet Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 0.5-1.3ml sodium citrate sample taken depending on infant weight
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infants with concern regarding late onset sepsis: Infants who are being investigated for late onset sepsis will be included. These infants may ultimately be classified in a number of ways, including culture positive late onset sepsis, culture negative late onset sepsis, necrotising enterocolitis or non infectious etiologies suspected (i.e prematurity)
  Interventions: Diagnostic Test: Platelet/Endothelial proteomics

INTERVENTIONS:
Diagnostic Test: Platelet/Endothelial proteomics — Samples taken will undergo a targeted proteomic investigation examining platelet/endothelial markers and associated extracellular vesicles

SUMMARY:
The PARENT study will examine platelet and endothelial associated proteins in preterm infants being investigated for late onset sepsis (LOS) to see if infants with fulminant sepsis can be prospectively identified using these markers

DETAILED DESCRIPTION:
Infants who are less than 34 weeks corrected gestational age at time of birth will be enrolled prior to any late onset sepsis investigations. At point of clinical concern for the development of late onset sepsis a 0.5-1.3ml sodium citrate sample will be taken. A targeted proteomic analysis using mass spectroscopy and flow cytometry will be performed and compared with the clinical diagnosis of the infant to examine if this can be used prospectively to identify infants with late onset sepsis

ELIGIBILITY:
Inclusion Criteria:

* <34 weeks corrected gestational age at birth
* Under investigation for Late Onset Neonatal Sepsis (Sepsis of onset >72 hours of age)

Exclusion Criteria:

* Major congenital anomaly
* Suspicion of an underlying haematological disorder affecting platelets
* Have received a platelet transfusion prior to sampling

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants less than 34 weeks corrected gestational age at birth who are undergoing investigations for late onset sepsis
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
A difference exists between infants with culture proven late onset sepsis and those without in platelet and endothelial proteomic profiles | 3 years
  Proteomic profiles including extracellular vesicles will be compared between those with and without culture proven sepsis

SECONDARY OUTCOMES:
To examine platelet markers in this same cohort and determine if they can distinguish between culture negative sepsis and non-sepsis | 3 years
  Proteomic profiles including extracellular vesicles will be compared between those with no culture proven sepsis and those without concern for sepsis/ a likely non infectious etiology
To determine if platelet activation markers correlate with severity of illness as established by prospective use of validated clinical scoring systems ( the novel neonatal Sequential organ failure assessment) | 3 years
  Proteomic profiles including extracellular vesicles will be compared with the nSOFA to examine if fulminant sepsis (Culture proven/Culture negative) can be predicted
To determine if platelet activation markers predict the development of necrotising enterocolitis (Radiological/Surgical) | 3 years
  Proteomic profiles including extracellular vesicles will be compared between those with and without radiological/surgical necrotising enterocolitis as final diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Maguire, Principal Investigator — University College Dublin
Locations (2):
- Ireland (2):
  - The National Maternity Hospital, Dublin, Dublin
  - The Rotunda Hospital, Dublin

IPD SHARING:
Plan to Share IPD: Undecided
Summary data will be available to other researchers, individual data will be withheld as much as required by GDPR requirements

REFERENCES:
- [Background] O'Reilly D, Murphy CA, Moore CM, Ni Ainle F, Gormley IC, Morrell CN, Curley A, Mc Callion N, Maguire P. Markers of platelet activation foR identification of late onset sEpsis in infaNTs: PARENT study protocol. Pediatr Res. 2024 Feb;95(3):852-856. doi: 10.1038/s41390-023-02812-x. Epub 2023 Sep 27. PMID 37758864